CLINICAL TRIAL: NCT05662683
Title: The Effect of Virtual Reality and Distraction Cards on Pain, Anxiety and Satisfaction Levels of Women Who Have Pap-Smears
Brief Title: The Effect of Virtual Reality and Distraction Cards on Pain
Acronym: Pap-Smear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate (Other Government)
Responsible Party: Principal Investigator, Mine Gokduman Keles, Midwifery, Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TurkishHKahramanmarasPH
Record Dates: First submitted 2022-11-15; First posted 2022-12-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Smear Layer; Cervical Cancer
Keywords: Virtual Reality; Distraction Cards; Pain; Anxiety; pap-smear
MeSH Terms: conditions — Smear Layer; Uterine Cervical Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: IT WILL BE APPLIED BY THE SAME HEALTH PERSONNEL WORKING AT THE KETEM CENTER After the women who meet the sample criteria of the study are determined and they accept to participate in the study, it will be determined which group the women are in from the list determined by randomization (determined from the www.randomizer.org site) according to the acceptance sequence number of the women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Working Group 1 (Experimental): From the preparation stage of the PAP-SMEAR removal procedure to the completion of the PAP-SMEAR removal procedure until the completion of the PAP-SMEAR removal procedure, after providing an internet connection with a smartphone for the image, clicking the youtube.com link and watching Relaxation (https://www.youtube.com/watch?v=H1iboKia3AQ) nature video virtual reality Goggles will be provided.
  Virtual reality glasses to be used in the research are not a medical device.
  Interventions: Other: Virtual Reality (VR)
- Working Group 2 (Experimental): Distraction cards containing five optical illusion figures will be shown to the women by the researcher
  Interventions: Other: Distraction Cards Practice Group
- Working Group 3 (Experimental): From the preparation stage of the PAP-SMEAR ALDIRAN procedure to the completion of the application process that takes PAP-SMEAR, the virtual reality glasses for breathing exercise by clicking the youtube.com link (https://www.youtube.com/watch?v=Pddb09FAs68) after providing an internet connection with a smartphone for the image. will be provided.
  Interventions: Other: Virtual Reality (VR) Breathing Exercise Group
- Control Group (No Intervention): The maintenance and applications in the routine PAP-SMEAR application will be done exactly.

INTERVENTIONS:
Other: Virtual Reality (VR) — Virtual reality glasses to be used in the research are not a medical device. This device is a technological glasses that works with compatible smartphones. During the PAP-SMEAR application to be made with this device, watching a nature video with VR is within the framework of midwifery care applications and is not a treatment option for any treatment method, agent or disease. Although the video watched with VR has no effect on medical treatment and care within the framework of midwifery care, it does not have any harmful effects on women. The participant can withdraw from this study at any time without giving any reason.
  Arms: Working Group 1
Other: Distraction Cards Practice Group — It will take about 3-5 minutes to show the cards. The selection of the cards to be used is based on the cards suggested in the literature.
  Arms: Working Group 2
Other: Virtual Reality (VR) Breathing Exercise Group — From the preparation stage of the PAP-SMEAR ALDIRAN procedure to the completion of the application process that takes PAP-SMEAR, the virtual reality glasses for breathing exercise by clicking the youtube.com link (https://www.youtube.com/watch?v=Pddb09FAs68) after providing an internet connection with a smartphone for the image. will be provided.
  Arms: Working Group 3

SUMMARY:
When the literature is examined, it is seen that virtual reality and distraction cards are used during medical procedures, and they have a reducing effect on pain perception and lowering the level of anxiety . On the other hand, no study has been found in the literature on the application of virtual glasses and distraction cards to women in the PAP-SMEAR process. However, in accordance with the results of the study conducted with the application of virtual reality glasses and distraction cards, it is thought that the application of virtual glasses will have a positive effect on reducing the perceived pain of women in the PAP-SMEAR process of distraction cards.

DETAILED DESCRIPTION:
Cervical cancer is the fourth most common cancer worldwide. Cervical cancer is one of the most successfully treatable types of cancer, as long as it is detected early and managed effectively. WHO recommends the use of PAP-SMEAR and HPV DNA primary screening test to prevent cervical cancer in women. . The crude incidence of cervical cancer per 100,000 women in Turkey in 2020 is . WHO has targeted a threshold of 4 per 100,000 women by 2030 for countries to eliminate cervical cancer. To achieve this goal, 90% of girls should be vaccinated with HPV until the age of 15, and 70% of women should be screened with high performance PAP-SMEAR and HPV DNA at the age of 35 and 45 For this reason, it is seen that the PAP-SMEAR test has an important place in the protection of women's health. For the Pap-Smear test procedure, gynecological examination and speculum examination are included . Experiencing pain, anxiety, shyness and fear during gynecological examination are among the barriers to applying for and taking the pap-smear test, which has an important place in protecting women's health In the literature, it is seen that virtual reality glasses and distraction cards, which are cognitive behavioral techniques, are used during medical procedures and have a reducing effect on the perception of pain and reduce the level of anxiety . No study has been found that examines the effect on satisfaction and satisfaction levels. However, in line with the results of the study, it is thought that the PAP-SMEAR procedure will have a positive effect on women's perceived pain and anxiety, and increase their satisfaction levels. It emphasizes the need for cost-effective and feasible non-pharmacological methods by healthcare professionals during PAP-SMEAR application.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years old, To see menstruation on the day of the operation, Turkish literate, No history of cervical surgery No active mental illness Did not use any pain or anxiety medication prior to the insertion procedure

Exclusion Criteria:

* Those with visual and auditory disabilities, Using misoprostol during the procedure, Using pain medication before the procedure

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It is seen that the PAP-SMEAR test has an important place in the protection of women's health. For the Pap-Smear test procedure, gynecological examination and speculum examination are included.
Enrollment: 132 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | (1) before inspection (2) speculum insertion (3) also performing the PAP-SMEAR import process; (4) will be evaluated after the end of the transaction.
  In the numerical evaluation scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
Verbal Category Scale | before inspection pap smear
  The Verbal Category Scale is also called the Simple Descriptive Scale, and this scale is based on the patient's choice of the most appropriate word to describe the pain condition. Pain severity ranges from mild to unbearable. In this scale, he used the words "mild", "disturbing", "severe", "very severe", "unbearable" to describe the severity of pain (Annex-4). The individual is asked to choose the appropriate category for his situation.
Verbal Category Scale | (1) before inspection (2) speculum insertion (3) also performing the PAP-SMEAR import process; (4) will be evaluated after the end of the transaction.
  The Verbal Category Scale is also called the Simple Descriptive Scale, and this scale is based on the patient's choice of the most appropriate word to describe the pain condition. Pain severity ranges from mild to unbearable. In this scale, he used the words "mild", "disturbing", "severe", "very severe", "unbearable" to describe the severity of pain (Annex-4). The individual is asked to choose the appropriate category for his situation.
State Anxiety Scale | before PAP-SMEAR procedure
  In the State Anxiety Scale; There are ten reversed statements, items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. When scoring, the reversed and direct statements are summed. Responses with a value of 4 indicate high anxiety in direct statements. In reversed expressions; Responses with a value of 1 indicate high anxiety, and responses with a value of 4 indicate low anxiety. The State Anxiety Scale score is calculated by adding 50 points to the difference between the total weighted scores of the reverse statements and the direct statements. Scoring in the State Anxiety Scale varies between 20-80 points. A score of less than 36 is considered no anxiety, a score of 37-42 is considered mild anxiety, and a score of 42 and above is considered high anxiety.
State Anxiety Scale | after PAP-SMEAR procedure
  In the State Anxiety Scale; There are ten reversed statements, items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. When scoring, the reversed and direct statements are summed. Responses with a value of 4 indicate high anxiety in direct statements. In reversed expressions; Responses with a value of 1 indicate high anxiety, and responses with a value of 4 indicate low anxiety. The State Anxiety Scale score is calculated by adding 50 points to the difference between the total weighted scores of the reverse statements and the direct statements. Scoring in the State Anxiety Scale varies between 20-80 points. A score of less than 36 is considered no anxiety, a score of 37-42 is considered mild anxiety, and a score of 42 and above is considered high anxiety.
Newcastle Nursing Care Satisfaction Scale | After PAP-SMEAR ALDIRAN procedure
  The scale is a 5-point Likert-type scale consisting of 19 items including nursing care. All items of the Newcastle Nursing Care Satisfaction Scale are positive. In the scoring used to determine the degree of satisfaction, there are statements such as "Not at all Satisfied=1 point, Slightly Satisfied=2 points, Fairly Satisfied=3 points, Very Satisfied=4 points, Extremely Satisfied=5 points". The scores given to the questions of all items marked on the score evaluation scale are added together. The maximum score obtained from the scale is 95, and the minimum score is 19. Evaluation is made by converting the total score obtained from the scale to 100. The increase in the total score obtained from the scale indicates that the patients' satisfaction with nursing is high.
Pulse Rate and Oxygen Saturation | 20 minutes during pap smear
  The pulse rate and saturation values of women will be evaluated physiologically using the sensor compatible planet 50n LT model pulse oximeter (Nellcor COVIDIEN SPO 2) device

CONTACTS AND LOCATIONS:
Overall Officials: mine gökduman keleş, Midwifery, Principal Investigator — Ministry of Health
Locations (1):
- TurkishMoHKahramanmarasPH, Kahramanmaraş, Turkey (Türkiye)

REFERENCES:
- [Background] Aktas D, Kumas MB, Odabasioglu BS, Kaya A. Effect of a Special Examination Gown and Nature-Based Sounds on Anxiety in Women Undergoing a Gynecological Examination. Clin Nurs Res. 2018 Jun;27(5):521-539. doi: 10.1177/1054773816686475. Epub 2017 Jan 8. PMID 28067068
- [Background] Angioli R, De Cicco Nardone C, Plotti F, Cafa EV, Dugo N, Damiani P, Ricciardi R, Linciano F, Terranova C. Use of music to reduce anxiety during office hysteroscopy: prospective randomized trial. J Minim Invasive Gynecol. 2014 May-Jun;21(3):454-9. doi: 10.1016/j.jmig.2013.07.020. Epub 2013 Aug 17. PMID 23962572
- [Background] Ulker K, Kivrak Y. The Effect of Information About Gynecological Examination on the Anxiety Level of Women Applying to Gynecology Clinics: A Prospective, Randomized, Controlled Study. Iran Red Crescent Med J. 2016 Feb 6;18(6):e23864. doi: 10.5812/ircmj.23864. eCollection 2016 Jun. PMID 27621913
- [Background] Basak T, Duman S, Demirtas A. Distraction-based relief of pain associated with peripheral intravenous catheterisation in adults: a randomised controlled trial. J Clin Nurs. 2020 Mar;29(5-6):770-777. doi: 10.1111/jocn.15131. Epub 2019 Dec 16. PMID 31793099
- [Background] Gupta A, Scott K, Dukewich M. Innovative Technology Using Virtual Reality in the Treatment of Pain: Does It Reduce Pain via Distraction, or Is There More to It? Pain Med. 2018 Jan 1;19(1):151-159. doi: 10.1093/pm/pnx109. PMID 29025113
- [Background] Gur EY, Apay SE. The effect of cognitive behavioral techniques using virtual reality on birth pain: a randomized controlled trial. Midwifery. 2020 Dec;91:102856. doi: 10.1016/j.midw.2020.102856. Epub 2020 Sep 28. PMID 33478718
- [Background] Hylton J, Milton S, Sima AP, Karjane NW. Cold Compress for Intrauterine Device Insertional Pain: A Randomized Control Trial. Womens Health Rep (New Rochelle). 2020 Aug 4;1(1):227-231. doi: 10.1089/whr.2020.0056. eCollection 2020. PMID 33786484
- See also: WHO. Cervical Cancer Country Profiles. 2021. — https://www.who.int/teams/noncommunicable-diseases/surveillance/data/cervical-cancer-profiles
- Available data/document: REVIEW: Journal of Continuing Medical — https://dergipark.org.tr/en/pub/sted/issue/52715/466811 — Ozturk, Y. (2020). Barriers to Women Having Pap Smear Screening Test .29 (1), 61-68. DOI: 10.17942/sted.466811